CLINICAL TRIAL: NCT05204810
Title: Optimisation of Anticoagulation in Patients on Nocturnal Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UGent_ClotNight
Record Dates: First submitted 2021-12-09; First posted 2022-01-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2021-12

CONDITIONS: Hemodialysis; Coagulation
Keywords: Hemodialyzer; Fibre Clotting; Nocturnal dialysis
MeSH Terms: conditions — Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Night_1dosis (Experimental): * anticoagulation at dialysis start
  * blood sampling 5min after start dosis, and at 1h, 4h and 8h after dialysis start
  * microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Other: Anticoagulation strategy; Other: Blood sampling; Other: Scanning of hemodialyzer with micro-computed tomography
- Night_2doses (Experimental): * anticoagulation split over dialysis start and halfway dialysis (after 4h)
  * blood sampling 5min after start dosis, and at 1h, 4h (1 sample before and 1 sample after the extra anticoagulant dosis) and 8h after dialysis start
  * microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Other: Anticoagulation strategy; Other: Blood sampling; Other: Scanning of hemodialyzer with micro-computed tomography

INTERVENTIONS:
Other: Anticoagulation strategy — For each session of this cross-over study, a different anticoagulation therapy is used: either 1 dose of anticoagulant or 2 doses of anticoagulant
Other: Blood sampling — During the study sessions, blood sampling is performed from the arterial blood line at different time points (5min, 60min, 240min and at the dialysis end)
Other: Scanning of hemodialyzer with micro-computed tomography — After the study sessions, the used hemodialyzers are scanned using a gold standard micro computed tomography technique.

SUMMARY:
To avoid clotting during extracorporeal treatment, an anticoagulant is added to the circuit, resulting in an increased risk for bleeding complications. In addition, there is evidence that a substantial number of fibers can become blocked before this is reflected in routinely observed parameters, or in termination of the dialysis session.

In standard hemodialysis of 4 hours, the anticoagulant is administered at the beginning of dialysis. For nocturnal hemodialysis, there is no hard evidence whether anticoagulation should be administered only at the dialysis start or with an extra dosing halfway the dialysis session.

The aim of this randomized cross-over study is to objectively quantify the number of patent fibers after nocturnal dialysis in two different settings: anticoagulation only at the dialysis start, and anticoagulation divided over two time points, i.e. dialysis start and halfway dialysis.

DETAILED DESCRIPTION:
This single centre, randomized cross-over study includes twenty stable chronic nocturnal hemodialysis patients with no coagulation disorder, active inflammation or chronic cumarin-derived medication.

Patients are randomized over 2 study arms. Each patient is dialyzed over 480min (at midweek) with 2 different settings: anticoagulation only at the dialysis start, and anticoagulation divided over two time points, i.e. dialysis start and halfway dialysis.

For each patient, the dialyzer, the dialysis mode (hemodialysis or hemodiafiltration) and the dialysis settings (blood flow, dialysate flow and substitution flow) are those as currently used by the patient during in-centre nocturnal dialysis.

To determine antiXa, blood samples are taken from the inlet dialysis line at the dialysis start (i.e. 5min after administration of the anticoagulant) and at 1h, 4h and 8h after dialysis start. During the session with 2 anticoagulant administrations, an extra blood sample is taken before as well as after the second anticoagulant administration.

Before the first test session, 1 blood sample is taken to determine antithrombin-III (AT-III).

In order to quantify dialyzer performance in terms of number of patent fibers, dialyzers are scanned after dialysis, using a glod standard non-invasive micro-CT technique.

Therefore, at the end of the dialysis session, a standard rinsing procedure of the hemodialyzer is performed using exact 300mL rinsing solution. Next, the hemodialyzer is dried using continuous positive pressure ventilation. Dialyzer fibre blocking is visualized in the dialyzer outlet potting using a 3D CT scanning technique on micrometer resolution. HECTOR is a High Energy CT scanner Optimized for Research, built by the Ghent University Centre for X-ray Tomography (UGCT) in collaboration with the UGCT spin-off company XRE (Gent, Belgium). In front of the X-ray source, the dialyzer is mounted vertically on a precision rotation stage, and radiographies were recorded over 360° with an angular interval of 0.15°. Scan conditions are optimized to maximize the signal-to-noise ratio based on the sample size and structure, and the scanner properties. The tube voltage is set at 80kV, at a power of 20 Watts, the maximal power that allowed imaging at a resolution of 25μm. A total of 2401 projections are recorded with 500ms exposure each, resulting in a total exposure time of 20 minutes. Acquired images at 0 (projection 1) and 360° (projection 2401) are compared to exclude movement of the hemodialyzer during the scanning process. Reconstruction of the raw projection data is performed with the Octopus Reconstruction software package, licensed by XRE23.

The non-blocked fibers are counted in the central cross-section of the dialyzer outlet potting in a computer-based way using the Fiji image processing toolkit of ImageJ analysis software (ImageJ 1.51H, NIH, Bethesda, USA), an open-source platform for biological-image analysis. By comparing the number of non-blocked fibers in used versus non-used dialyzers, the percentage of fiber blocking can be calculated.

By comparing the number of open fibers between the 2 test sessions (1 versus 2 anticoagulant administrations), the difference can objectively be scored for prolonged (nocturnal) dialysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* experienced stable dialysis sessions during the last 4 weeks
* nocturnal in-centre hemodialysis
* well functioning vascular access

Exclusion Criteria:

* known coagulation disorder
* active inflammation
* malignancy
* no coumarin-derived medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of open fibers in hemodialyzer | 2 weeks
  By scanning the hemodialyzers post dialysis using a reference micro-CT scanning technique, images are obtained from dialyzer cross-sections. Black dots can be counted as open fiber. By counting the number of open fibers and relating this number with the total numerb of fibers in sterile dialyzers, the percentage of open fibers can be quantified.

SECONDARY OUTCOMES:
Absolute value and change of the clotting parameter antiXa at different time points during dialysis | 2 weeks
  AntiXa (i.e. a measure to indicate anticoagulation by low molecular weight heparins) is followed in the patient at dialysis start and after 1, 4, and 8h.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, Prof dr, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital - Nephrology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No